CLINICAL TRIAL: NCT00910091
Title: A Phase II International Multicentre Randomised Open Label Study of Oral Steroid Sulphatase Inhibitor BN83495 Versus Megestrol Acetate (MA) in Women With Advanced or Recurrent Endometrial Cancer
Brief Title: The Study of Oral Steroid Sulphatase Inhibitor BN83495 Versus Megestrol Acetate (MA) in Women With Advanced or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X-55-58064-004; 2009-010613-68 (EudraCT Number)
Record Dates: First submitted 2009-05-21; First posted 2009-05-29 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Antitumour efficacy in women with advanced endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — irosustat; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A- BN 83495- 40mg (Experimental): After eligibility is confirmed, subjects will be randomised at baseline. The randomisation number and associated treatment for the total study will be allocated by an Interactive Voice Response System (IVRS) service
  Interventions: Drug: BN83495
- B- MA - 160mg (Active Comparator): After eligibility is confirmed, subjects will be randomised at baseline. The randomisation number and associated treatment for the total study will be allocated by an Interactive Voice Response System (IVRS) service
  Interventions: Drug: Megestrol Acetate (MA)

INTERVENTIONS:
Drug: BN83495 — BN83495 will be administered as a 40 mg tablet once a day orally
  Arms: A- BN 83495- 40mg
Drug: Megestrol Acetate (MA) — MA will be administered orally as 160mg daily
  Arms: B- MA - 160mg

SUMMARY:
This trial will explore the safety and efficacy of BN83485 compared to Megestrol Acetate (MA) on progression free survival (PFS) in post menopausal patients with endometrial cancer.

DETAILED DESCRIPTION:
The Primary Objective in this study is to determine the antitumour efficacy of BN83495 measured by the percentage of women with advanced or recurrent endometrial cancer who have neither progressed nor died after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures
* Post-menopausal or ovariectomised female patients over the age of 18 years with advanced or recurrent endometrial carcinoma
* Histologically confirmed diagnosis endometrial carcinoma (primary tumour or metastasis)
* Not eligible for surgery or radiotherapy alone, at Investigator's discretion
* Documented Estrogen Receptor (ER) positivity in the primary tumour or in the metastatic tissue if the primary tumour is unavailable (ER positivity is defined by at least 10% positive cells)
* No other history of malignant disease except treated basal cell or in situ cervical carcinoma in the previous 5 years. In case of previous malignant disease, pathological confirmation of metastatic endometrial cancer will be done at Investigator's discretion
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤2
* At least one measurable disease site

  * minimum indicator lesion size: 20 mm (conventional techniques) or 10 mm (spiral CT scan)
  * target lesions not situated in irradiated area
* Life expectancy ≥6 months
* Adequate organ function as defined by the following criteria:

  * Haemoglobin ≥10 g/dL
  * Absolute neutrophil count (ANC) ≥1500/μL
  * Platelets ≥100,000/μL
  * Serum creatinine ≤1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥50 ml/min
  * Serum AST and serum ALT ≤2.5x ULN or AST and ALT ≤5x ULN if liver metastases
  * Total serum bilirubin ≤1.5x ULN
  * Serum albumin ≥3.0 g/dL
  * Cardiac function ≤New York Heart Association (NYHA) class II
* Patients must have recovered from surgery, radiotherapy and toxicities of adjuvant chemotherapy treatment if applicable
* Patients must be willing and able to participate in a clinical trial (including the completion of all necessary study procedures)
* Patients must be able to swallow oral medication

Exclusion Criteria:

* Use of any investigational agent in the 4 weeks prior to enrollment in this study
* Prior systemic treatment for endometrial cancer (including hormonal treatment, chemotherapy, antiangiogenic or targeted therapies)with the exception of chemotherapy in the adjuvant setting, having been completed at least 6 months prior to randomisation
* Known central nervous system (CNS) metastases
* Ongoing cardiac dysrhythmias of National Cancer Institute Common Toxicity Criteria Adverse Events (NCI CTC AE) grade ≥2, atrial fibrillation of any grade, QTcF interval >460 msec.
* Patients with contraindications to Megestrol Acetate (MA) including hypersensitivity to one of the drug product, any active arterial or venous thromboembolic event and/or uncontrolled hypertension. Patients receiving anticoagulation for a prior thromboembolic event may be enrolled in the study at the Investigator's discretion
* Concomitant use of carbonic anhydrase II inhibitors (e.g. acetazolamide, dichlorphenamide, methazolamide)
* History of hypersensitivity to BN83495 or drugs with a similar chemical structure
* Likely to require treatment during the study with drugs that are not permitted by the study protocol
* Abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the patient's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (54):
- Belgium (4):
  - Onze-Lieve-Vrouwzickenhuis-Campus Aalst, Aalst
  - Centre Jules Bordet, Brussels
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - Sint Augustinus, Wilrijk
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Gynekologicko-porodnicka klinika, Prague
  - Krajska zdravotni s.r.o. - Masarykova nemocnice Usti nad Labem, Ústí nad Labem
- France (14):
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre René Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Hungary (2):
  - BAZ Megyei Kórház és Egyetemi Oktató Kórház, Sugártherápiás és Onkológiai Intézet, Miskolc
  - Szegedi Tudományegyetem Szent-Györgyi Albert Orvos-és Gyógyszerésztudományi Centrum, Szeged
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - Piejuras Hospital, Oncologic Clinic, Liepāja
  - Riga Eastern CUH - Latvian Oncology Centre, Department No 9, Riga
- Lithuania (2):
  - Kauno universiteto medicinos kliniku onkologijos ligonine, Kaunas
  - Vilniaus universiteto Onkologijos institutas, Vilnius
- Institutul Oncologic, Chisinau, Moldova
- Poland (4):
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Uniwersytet Medyczny, Poznan
  - Oddział Ginekologii Onkologicznej Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im Karola Marcinkowskiego w Poznaniu, Poznan
  - Centrum Onkologii Instytut Marii Sklodowskiej Curie, Warsaw
- Russia (8):
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - Medical Radiology Research Center of RAMS, Obninsk
  - GUZ "Orenburg Regional Clinical Oncology Dispensary", Orenburg
  - Perm Regional Oncology Dispensary, Perm
  - GUZ of Stavropol Territorial Clinical Oncological Dispensary, Pyatigorsk Branch, Pyatigorsk
  - FGU "Research Institute of Oncology named after N.N.Petrov", Saint Petersburg
  - Saint-Petersburg GUZ City Clinical Oncology Dispensary, Saint Petersburg
  - OOO "Sibmedcenter", Tomsk
- Spain (4):
  - H. Universitario Vall d´Hebron, Barcelona
  - H. Universitario 12 de Octubre, Madrid
  - H. Universitario Central de Asturias, Oviedo
  - H. Clinico Universitario San Carlos, San Carlos
- Ukraine (4):
  - Oblasnyi onkologichnyi klinichnyi dyspanser, misto Uzhgorod. Uzhgorods'kyi natsionalnyi universytet, Chernivtsi
  - DU "Instytut medychnoi radiologii im. S.P. Grygorieva AMN Ukrainy", Kharkiv
  - DU "Natsionalnyi instytut raku", m. Kyiv, Kyiv
  - Lvivskyi derzhavnyi onkologichnyi regionalnyi likuvalno-diagnostychnyi tsentr, Lviv
- United Kingdom (5):
  - Beatson Oncology Centre, Gartnavel General Hospital, Glasgow
  - St James's University Hospital, Leeds
  - University Hospitals of Leicester, Leicester Royal Infirmary, Leicester
  - University of Liverpool Clatterbridge Centre for Oncology, Liverpool
  - Christie Hospital NHS Trust, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: BN83495 40 mg: BN83495 (Irosustat) 40 mg tablet by mouth once daily
- Arm B: MA 160 mg: Megestrol Acetate (MA) 160 mg tablet by mouth once daily
Period: Pre-assignment
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Started | 36 | 37
Completed | 36 | 35
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Treatment and Survival
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Started | 36 | 35
Completed | 32 | 31
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B: MA 160 mg: MA 160 mg tablet by mouth once daily
- Total: Total of all reporting groups
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Median (Standard Deviation); unit: Years] | 68.1 (11.4) | 67.4 (8.6) | 67.7 (10.0)
Age, Customized [Number; unit: Participants]
  18-64 years | 12 | 16 | 28
  65-75 years | 13 | 15 | 28
  >75 years | 11 | 6 | 17
Sex/Gender, Customized [Number; unit: Participants]
  Female | 36 | 37 | 73
Region of Enrollment [Number; unit: Participants]
  France | 8 | 7 | 15
  United Kingdom | 7 | 7 | 14
  Belgium | 6 | 2 | 8
  Russian Federation | 6 | 8 | 14
  Czech Republic | 3 | 5 | 8
  Poland | 2 | 2 | 4
  Ukraine | 2 | 2 | 4
  Lithuania | 1 | 1 | 2
  Spain | 1 | 1 | 2
  Latvia | 0 | 1 | 1
  Moldova, Republic of | 0 | 1 | 1
BMI (Body Mass Index) [Number; unit: Participants]
  <18.5 kg/m2 | 1 | 0 | 1
  18.5 - 25 kg/m2 | 10 | 10 | 20
  >25 - 30 kg/m2 | 10 | 8 | 18
  >30 kg/m2 | 12 | 17 | 29
  Missing | 3 | 2 | 5
Race [Number; unit: Subjects]
  Black / African American | 0 | 1 | 1
  Caucasian / White | 36 | 36 | 72
Eastern Cooperative Oncology Group(ECOG) Performance Status Score [Mean (Standard Deviation); unit: Units on a scale] — ECOG score ranges from 0 to 5, where 0: Asymptomatic, 1: Symptomatic but completely ambulatory, 2: Symptomatic (<50% in bed during the day - ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours), 3: Symptomatic (>50% in bed, but not bedbound - capable of only limited self-care, confined to bed or chair 50% or more of waking hours), 4: Bedbound (Completely disabled- cannot carry on any self-care) and 5: Death.
  Units on a scale | 0.8 (0.6) | 0.7 (0.7) | 0.7 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Advanced or Recurrent Endometrial Cancer Who Have Neither Progressed Nor Died
Description: Subject continuation in the study and Response Evaluation Criteria in Solid Tumours (RECIST) assessment has been based on investigator assessment and not on central review. The 6 month timepoint is defined as the treatment start date +183 days (26 weeks).
Time Frame: Up to 6 months
Population: Intent-to-treat (ITT) population includes all randomized subjects who received at least one dose of study medication.
Measure: Number (90% Confidence Interval); unit: Percentage of subjects
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 37
Percentage of subjects | 36.1 [24.3 to 49.8] | 54.1 [40.8 to 66.8]

2. Secondary Outcome: Percentage of Participants With Adverse Event (AE)
Description: Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life threatening/disabling and Grade 5: Death
Time Frame: Up to Day 28 follow-up
Population: Safety Population: All randomised subjects who received at least one dose of study medication.
Measure: Number; unit: Percentage of subjects
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 35
Percentage of subjects
  Any AEs | 88.9 | 82.9
  Any Treatment Emergent AEs (TEAEs) | 88.9 | 82.9
  Intensity of TEAEs - Grade 5 | 2.8 | 2.9
  Intensity of TEAEs - Grade 4 | 5.6 | 0.0
  Intensity of TEAEs - Grade 3 | 22.2 | 25.7
  Intensity of TEAEs - Grade 2 | 63.9 | 45.7
  Intensity of TEAEs - Grade 1 | 80.6 | 74.3
  Intensity of TEAEs - Missing | 5.6 | 0.0
  Causality of TEAEs - Related | 55.6 | 37.1
  Causality of TEAEs - Not related | 77.8 | 77.1
  TEAEs Leading to Withdrawal | 8.3 | 2.9
  TEAEs Leading to Death | 2.8 | 2.9
  Serious Adverse Events (SAEs) | 25.0 | 17.1

3. Secondary Outcome: Tolerability of BN83495 Based on Length of Exposure
Description: Length of exposure includes interruptions.
Time Frame: Up to 2 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Week
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 35
Week | 34.94 (38.85) | 55.20 (49.48)

4. Secondary Outcome: Tolerability of BN83495 Based on Cumulative Dose Administered
Description: Cumulative dose is the actual total dose administered.
Time Frame: Up to 2 years
Population: Safety Population
  Missing number of subjects = 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 33
mg | 9452.22 (10799.16) | 60703.03 (51726.14)

5. Secondary Outcome: Tolerability of BN83495 Based on Dose Interruptions and Reason for Interruptions
Description: Percentage of participants who had dose interruptions and reason for interruptions as AE, study treatment forgotten, and other reasons.
Time Frame: Up to 2 years
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 35
Percentage of participants
  Dose Interruptions | 27.8 | 34.5
  Reason for Interruptions (AE) | 16.7 | 8.6
  Reason for Interruptions (Treatment forgotten) | 0.0 | 8.6
  Reason for Interruptions (Other) | 13.9 | 20.0

6. Secondary Outcome: Percentage of Participants >65 Years of Age With No Change or Deterioration, Improvement of <10%, or Improvement of ≥10% on the EuroQoL Score
Description: EuroQoL (Quality of Life)-5 Dimensions (EQ-5D) is a participant answered questionnaire scoring 5 dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.
Time Frame: Up to week 32
Population: ITT population.
  Three subjects withdrawn the consent from MA 160 mg group and did not have EuroQoL score up to week 32.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 24 | 18
Percentage of participants
  No Change or Deterioration at week 2 | 54.2 | 50.0
  No Change or Deterioration at week 4 | 54.2 | 61.1
  No Change or Deterioration at week 8 | 25.0 | 50.0
  No Change or Deterioration at week 16 | 25.0 | 50.0
  No Change or Deterioration at week 24 | 16.7 | 33.3
  No Change or Deterioration at week 32 | 16.7 | 22.2
  Improvement of <10% at week 2 | 0.0 | 5.6
  Improvement of <10% at week 4 | 4.2 | 5.6
  Improvement of <10% at week 8 | 4.2 | 5.6
  Improvement of <10% at week 16 | 0.0 | 0.0
  Improvement of <10% at week 24 | 0.0 | 5.6
  Improvement of <10% at week 32 | 8.3 | 5.6
  Improvement of ≥10% at week 2 | 20.8 | 5.6
  Improvement of ≥10% at week 4 | 16.7 | 16.7
  Improvement of ≥10% at week 8 | 16.7 | 16.7
  Improvement of ≥10% at week 16 | 12.5 | 5.6
  Improvement of ≥10% at week 24 | 12.5 | 5.6
  Improvement of ≥10% at week 32 | 0.0 | 5.6

7. Secondary Outcome: Percentage of Participants With Clinical Benefit [Including Completed Response (CR), Partial Response (PR), and Stable Disease (SD)] ≥12 Weeks
Description: CR: Disappearance of all known disease & no new sites / disease related symptoms confirmed at least 12 weeks after initial documentation. Disappearance of all non-target lesions. Normalization of tumor marker level confirmed at least 12 weeks after initial documentation.
  PR: Minimum 30% decrease in sum of the longest diameters of target lesions, taking as a reference the baseline sum of the longest diameters confirmed at least 12 weeks after initial documentation. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing. As well as persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above normal limits.
  RECIST defines SD for target lesions as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, no occurrence of progression disease for non-target lesions, and no new lesions.
Time Frame: Up to 2 years
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 37
Percentage of Participants | 13 (36.1) | 19 (51.4)
Statistical Analysis 1: Comparison: Arm A: BN83495 40 mg vs Arm B: MA 160 mg; Test type: Superiority or Other; p = 0.1895, Kaplan-Meier Analysis

8. Secondary Outcome: Percentage of Participants With Overall Response (OR) Including CR and PR
Time Frame: Up to 2 years
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 37
Percentage of Participants | 3 (8.3) | 11 (29.7)
Statistical Analysis 1: Comparison: Arm A: BN83495 40 mg vs Arm B: MA 160 mg; Test type: Superiority or Other; p = 0.0203, Kaplan-Meier Analysis

9. Secondary Outcome: Percentage of Participants With First Documentation of Objective Tumour Progression From Randomisation
Time Frame: Up to 2 years
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 37
Percentage of Participants | 30 (83.3) | 24 (64.9)

10. Secondary Outcome: Duration of Response (DR) in Responders
Description: DR is defined as period from the time that measurement criteria are first met for CR or PR until first date of documented Progressive Disease (PD) or death. DR was assessed in participants with a best overall response of CR or PR.
Time Frame: At 2 years
Population: ITT population.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 37
Weeks | NA [23.14 to NA] — NA = Values are not calculable | 105.14 [47.71 to NA] — NA = Values are not calculable
Statistical Analysis 1: Comparison: Arm A: BN83495 40 mg; Test type: Superiority or Other; p = 0.6980, Kaplan-Meier Analysis

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of enrollment to the date of death due to any cause.
Time Frame: At 2 years
Population: ITT population.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 37
Weeks | 63.43 [37.57 to 100.29] | NA [56.14 to NA] — NA = Values are not calculable
Statistical Analysis 1: Comparison: Arm A: BN83495 40 mg; Test type: Superiority or Other; p = 0.3078, Kaplan-Meier Analysis

12. Secondary Outcome: Progression Free Survival (PFS): Time From Randomisation Until Objective Tumour Progression or Death From Any Cause
Time Frame: Up to 2 years
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Arm A: BN83495 40 mg | Arm B: MA 160 mg
Number analyzed (Participants) | 36 | 37
Weeks | 16.14 [9.00 to 31.43] | 40.14 [16.29 to 64.00]
Statistical Analysis 1: Comparison: Arm A: BN83495 40 mg; Test type: Superiority or Other; p = 0.0484, Kaplan-Meier Analysis

ADVERSE EVENTS:
Time Frame: Up to Day 28 follow-up
Arm/Group | A- BN 83495- 40mg | B- MA - 160mg
Serious Adverse Events (participants affected / at risk) | 9/36 | 6/35
Other Adverse Events (participants affected / at risk) | 32/36 | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A- BN 83495- 40mg (N=36) | B- MA - 160mg (N=35)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A- BN 83495- 40mg (N=36) | B- MA - 160mg (N=35)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 14 (14) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 6 (6) | 2 (2)
Fatigue (General disorders) | 6 (6) | 4 (4)
Spinal Pain (General disorders) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 6 (6)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Blood Creatinine Increased (Investigations) | 3 (3) | 1 (1)
Blood Urea Increased (Investigations) | 2 (2) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Hot Flush (Vascular disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contrast Media Allergy (Immune system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No